CLINICAL TRIAL: NCT03849014
Title: Comparison of Biochemical Changes in Patients With Trochanteric Region Fracture Fixation With Dynamic Hip Screw Versus Proximal Femoral Nail
Brief Title: Comparison of Biochemical Changes in Patients With Trochanteric Region Fracture Fixation With DHS Versus PFN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kushtrim Grezda (Other)
Collaborators: University Clinical Centre of Kosova (Other)
Responsible Party: Sponsor-Investigator, Kushtrim Grezda, Principal Investigator, Clinical Research, University Clinical Centre of Kosova
Organization: University Clinical Centre of Kosova (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGrezda
Record Dates: First submitted 2019-01-17; First posted 2019-02-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Inflammatory response; Interleukin-6; Comparative study
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic Hip Screw (Active Comparator): Dynamic Hip Screw is used for internal fixation of fractures of the certain types of hip fractures. The implant assembly consisting of a lag screw, a side plate, and cortical screws that fix the side plate to the proximal femoral shaft.
  Interventions: Procedure: Dynamic Hip Screw
- Proximal Femoral Nail (Active Comparator): The Proximal Femoral Nail offers osteosynthesis for the several types of hip fractures. It consists of an anatomically curved nail, double neck screw, and two locking screws for distal end.
  Interventions: Procedure: Proximal Femoral Nail

INTERVENTIONS:
Procedure: Dynamic Hip Screw — Dynamic Hip Screw fixation: Fracture will be reduced under image intensifier. The incision will be made 7-10 cm with a lateral approach. The fascia lata will be incised and the vastus lateralis muscle will be splited along the axis of the femur, without stripping the periosteum. A135° angle guide will be inserted in the lower half of the femoral neck. The barrel of the plate will be guided to the hip screw by direct palpation to minimize the soft-tissue injury. After the insertion of the cortical screw, soft tissue will be protected with 4.5mm drill sleeve during drilling and tapping.
  Arms: Dynamic Hip Screw
Procedure: Proximal Femoral Nail — Proximal Femoral Nail fixation: Fracture will be reduced under image intensifier. The incision 2-3 cm with a lateral approach that extended from the cranial part to the tip of the greater trochanter. After palpating the greater trochanter tip, the nail will be then introduced manually into the femoral shaft. The guide wire of the anti-rotational hip blade then introduced. The hip blade should be introduced in the direction of the lower half of the femoral neck. Drilling will be performed under soft-tissue protection with a retractor. The blade will be inserted, and a distal static locking screw and end cap will be inserted under soft tissue protection with a drill sleeve.
  Arms: Proximal Femoral Nail

SUMMARY:
Hip fractures are one of the most frequent fractures in older adults. There is still controversy which surgical strategy is the best option for treatment of hip fractures especially trochanteric region fractures. Surgical intervention that follows hip fracture induces biochemical, physiological and fibrinolytic changes that are so-called "second hit phenomenon" which trigger systemic inflammatory response syndrome. The investigators are aiming to study this phenomenon after two different surgical procedures and help surgeons in everyday practice to choose the most suitable surgical treatment for patients with trochanteric region fracture and give the scientific community more evidence which methods is better since there is still controversy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trochanteric region fractures AO/OTA 31.A1-31.A2
* Time from fracture till surgery up to 1 week
* American Society of Anesthesiologists Classification (ASA) I-III
* Willing to participate

Exclusion Criteria:

* Polytrauma patients
* Open fractures
* Existing local or systemic infection
* Pre-existing coagulatory disorder
* Existing malignancy
* Corticosteroid use
* Systemic inflammatory disease
* Voluntary withdraws of the patient

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
The difference of the level of IL-6 in operated patients. | 1 hour before and 24 hours after operation
  The blood will be collected and after that centrifuged and then stored in -20 grade celsius. The analysis of each sample will be performed no later than 3 months.

SECONDARY OUTCOMES:
The difference of the level of CRP in operated patients. | 1 hour before and 24 hours after operation. Length of operation, length of incision, blood loss perioperatively. Complication and mortality rate within 1 month after OP
  The analysis will be performed immediately after the blood sample is collected.
The difference of the level of D-dimer | 1 hour before and 24 hours after operation
  The analysis will be performed immediately after the blood sample is collected.
The difference of the level of ESR | 1 hour before and 24 hours after operation
  The analysis will be performed immediately after the blood sample is collected.
The difference of the length of operation | Intra-operatively
  The stopwatch will be turned on from the incision until the end of the skin suture
The difference of the level of length of incision | After the wound closure
  The measure will be made with centimeters (cm)
Blood loss | Levels of HB before and after surgery. Also the total volume of blood transfusion.
  HB-balance method will be used
Complications after surgery | Within 1 month after surgery
  All complications that might occur after surgery will be registered
Mortality rate | Within 1 month after surgery
  The mortality of patients that might happen after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kushtrim Grezda, MD, Principal Investigator — University Clinical Centre of Kosova
Locations (1):
- Qendra Klinike Universitare e Kosoves, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided